CLINICAL TRIAL: NCT00975000
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Using Cinacalcet to Correct Hypercalcemia in Renal Transplant Recipients With Autonomous Hyperparathyroidism
Brief Title: Treatment of Autonomous Hyperparathyroidism in Post Renal Transplant Recipients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20062007
Record Dates: First submitted 2009-09-10; First posted 2009-09-11 (Estimated); Results first posted 2016-01-29 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-09

CONDITIONS: Chronic Allograft Nephropathy; Chronic Kidney Disease; Chronic Renal Failure; Disordered Mineral Metabolism; End Stage Renal Disease; Hyperparathyroidism; Hypophosphatemia; Kidney Disease; Kidney Transplantation; Post Renal Transplantation
Keywords: Intervention; Cinacalcet; Sensipar; Mimpara; hyperparathyroidism; calcium; osteodystrophy; hypercalcemia; renal; transplant; acute rejection; kidney transplant failure; hypophosphatemia
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic; Hyperparathyroidism; Hypophosphatemia; Kidney Diseases; Hypercalcemia | interventions — Cinacalcet

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cinacalcet (Experimental): Participants received cinacalcet at a starting dose of 30 mg orally once daily for 52 weeks. Cinacalcet dose was titrated every 4 weeks during the dose-titration phase and during study visits in the maintenance phase based on intact parthyroid hormone (iPTH) values, corrected total serum calcium values, and safety assessments.
  Interventions: Drug: Cinacalcet
- Placebo (Placebo Comparator): Participants received placebo orally once daily for 52 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cinacalcet — Possible sequential doses are 30, 60, 90, 120, and 180 mg.
  Other Names: Mimpara; Sensipar
  Arms: Cinacalcet
Drug: Placebo — Administered orally following the same dosing regimen as the experimental arm.
  Arms: Placebo

SUMMARY:
Hyperparathyroidism (HPT) is common in people with a kidney transplant. Patients with HPT often have high parathyroid hormone (PTH) levels and may have large parathyroid glands in the neck. Patients with HPT can develop bone disease (osteodystrophy). This bone disease can cause bone pain, fractures, and poor formation of red blood cells. Other problems from HPT may include increases in blood levels of calcium (hypercalcemia) and low blood levels of phosphorus (hypophosphatemia). The high calcium levels may cause calcium to deposit in body tissues. Calcium deposits can cause arthritis (joint pain and swelling), muscle inflammation, itching, gangrene (death of soft tissue), heart and lung problems or kidney transplant dysfunction (worsening of kidney transplant function). The purpose of this study is to evaluate the effects of cinacalcet (Sensipar/Mimpara) on high calcium levels in the blood in patients with HPT after a kidney transplant.

ELIGIBILITY:
Inclusion Criteria:

* Received a kidney transplant ≥ 9 weeks at time of Screening and ≤ 24 months before first dose
* May be the first kidney transplant or a repeat kidney transplant.
* Subjects with a functional, stable kidney transplant, defined as MDRD estimated glomerular filtration rate (eGFR) ≥ 30 mL/min/1.73 m² (chromic kidney disease stage 3 or better) at Screening.
* Men or women ≥ 18 years at the start of Screening (ie, time of informed consent).
* Corrected total serum calcium > 10.5 mg/dL (2.63 mmol/L), defined as the mean of 2 values in Screening period.
* iPTH > 100 pg/mL (10.6 pmol/L), during the Screening period (obtained at either Screen 1 or Screen 2).

Exclusion Criteria:

* Received cinacalcet therapy post-transplant for more than 14 days cumulatively post-transplant. If cinacalcet therapy was received for a total of 14 days or less post-transplant, there must be a 4-week washout before subject is eligible for screening (Note: This does not exclude pre-transplant use of cinacalcet).
* Anticipated parathyroidectomy within 6 to12 months after Randomization.
* Ongoing therapy with bisphosphonates or use within 6 months prior to Screening.
* Ongoing use of 1,25-dihydroxyvitamin D3 (including other active vitamin D metabolites or analogues) or use within 30 days prior to Screening.
* Ongoing use of calcium supplements or use within 30 days prior to Screening.
* Ongoing use of phosphate binders (calcium or non-calcium containing) or use within 30 days prior to Screening.
* Ongoing use of a thiazide diuretic.
* Subjects with a history of seizures who had a seizure within the 3 months prior to Randomization, which required adjustments to the seizure medication.
* Acute Kidney Injury (AKI) or renal biopsy within 6 weeks prior to Screening, unless it is an institutional protocol-driven biopsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2009-12-03 (Actual); Primary Completion 2012-09-13 (Actual); Study Completion 2013-04-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (50):
- United States (15):
  - Research Site, Phoenix, Arizona
  - Research Site, Tempe, Arizona
  - Research Site, San Francisco, California
  - Research Site, Aurora, Colorado
  - Research Site, Gainesville, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Evanston, Illinois
  - Research Site, Springfield, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, New York, New York
  - Research Site, Bethlehem, Pennsylvania
  - Research Site, Nashville, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
- Australia (4):
  - Research Site, Camperdown, New South Wales
  - Research Site, Westmead, New South Wales
  - Research Site, Woodville South, South Australia
  - Research Site, Parkville, Victoria
- Research Site, Vienna, Austria
- Belgium (3):
  - Research Site, Brussels
  - Research Site, Ghent
  - Research Site, Leuven
- Canada (5):
  - Research Site, Calgary, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, London, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
- France (5):
  - Research Site, Bordeaux
  - Research Site, Montpellier
  - Research Site, Nantes
  - Research Site, Paris
  - Research Site, Toulouse
- Germany (2):
  - Research Site, Berlin
  - Research Site, Kiel
- Italy (3):
  - Research Site, Genova
  - Research Site, Milan
  - Research Site, Padua
- Poland (5):
  - Research Site, Gdansk
  - Research Site, Katowice
  - Research Site, Lodz
  - Research Site, Poznan
  - Research Site, Szczecin
- Spain (4):
  - Research Site, MÃ¡laga, AndalucÃ-a
  - Research Site, Barcelona, CataluÃ±a
  - Research Site, L'Hospitalet de Llobregat, CataluÃ±a
  - Research Site, Madrid
- Switzerland (3):
  - Research Site, Bern
  - Research Site, Geneva
  - Research Site, Zurich

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 33 centers in 11 countries (Australia, Austria, Belgium, Canada, France, Germany, Italy, Poland, Spain, Switzerland, and USA).
  First patient enrolled on 15 October 2009 and last patient enrolled on 07 March 2012.
Pre-assignment Details: The study consisted of a 20-week titration phase, a 6-week efficacy assessment phase (EAP), a 26-week blinded maintenance phase and a 4-week follow-up phase. Randomization was stratified by corrected total serum calcium (Ca); enrollment into the low Ca stratum was limited to ≤70% of patients to ensure at least 30% enrollment in the high Ca stratum.
Groups:
- Cinacalcet: Participants received cinacalcet at a starting dose of 30 mg orally once daily for 52 weeks. Cinacalcet dose was titrated every 4 weeks during the dose-titration phase and during study visits in the maintenance phase based on intact parathyroid hormone (iPTH) values, corrected total serum calcium values, and safety assessments.
Period: Overall Study
Arm/Group | Placebo | Cinacalcet
Started | 57 | 57
Completed Titration Phase | 54 | 55
Completed Efficacy Assessment Phase | 54 | 54
Completed Maintenance Phase | 52 | 52
Completed | 52 (Completed post-treatment follow-up phase) | 52 (Completed post-treatment follow-up phase)
Not Completed | 5 | 5
Not completed — Other | 1 | 0
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol-specified Criteria | 1 | 0
Not completed — Non-compliance | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Cinacalcet: Participants received cinacalcet at a starting dose of 30 mg orally once daily for 52 weeks. Cinacalcet dose was titrated every 4 weeks during the dose-titration phase and during study visits in the maintenance phase based on the iPTH values, corrected total serum calcium values, and safety assessments.
- Total: Total of all reporting groups
Arm/Group | Placebo | Cinacalcet | Total
Number analyzed (Participants) | 57 | 57 | 114
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.7 (9.9) | 53.0 (10.7) | 52.3 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 26 | 51
  Male | 32 | 31 | 63
Race/Ethnicity, Customized [Number; unit: participants]
  White or Caucasian | 46 | 47 | 93
  Black or African American | 4 | 5 | 9
  Hispanic or Latino | 1 | 2 | 3
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Other | 1 | 1 | 2
Stratification Factor: Albumin-corrected Calcium Level [Number; unit: participants]
  Corrected calcium ≤ 11.2 mg/dL | 22 | 23 | 45
  Corrected calcium > 11.2 mg/dL | 35 | 34 | 69
Corrected Total Serum Calcium [Mean (Standard Deviation); unit: mg/dL] | 11.31 (0.50) | 11.28 (0.41) | 11.29 (0.45)
Intact Parathyroid Hormone [Mean (Standard Deviation); unit: pg/mL] | 307.5 (180.5) | 327.7 (262.6) | 317.6 (224.5)
Serum Phosphorus [Mean (Standard Deviation); unit: mg/dL] — Data available for 56 participants in each treatment group.
  mg/dL | 2.48 (0.52) | 2.66 (0.54) | 2.57 (0.54)
Estimated Glomerular Filtration Rate (eGFR) [Mean (Standard Deviation); unit: mL/min/1.73 m²] — eGFR was calculated using the Modification of Diet in Renal Disease (MDRD) formula.
  mL/min/1.73 m² | 54.68 (14.79) | 57.00 (17.31) | 55.84 (16.07)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Mean Corrected Total Serum Calcium Value < 10.2 mg/dL (2.55 mmol/L) During the Efficacy Assessment Phase (EAP)
Time Frame: Weeks 21 to 26 (EAP)
Population: Full analysis set (all randomized participants excluding participants determined to have graft failure prior to week 26)
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Cinacalcet
Number analyzed (Participants) | 57 | 57
percentage of participants | 3.5 | 78.9
Statistical Analysis 1: Comparison: Placebo vs Cinacalcet; The primary endpoint was tested at a significance level of 0.05; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test stratified by baseline corrected total serum calcium level (≤ 11.2 mg/dL and > 11.2 mg/dL); Chi-Square test statistic = 66.437
Statistical Analysis 2: Comparison: Placebo vs Cinacalcet; Test type: Superiority or Other; Odds Ratio (OR) = 91.41, 95% CI 2-sided [18.76 to 445.41] — Odds ratio of Cinacalcet/Placebo
Statistical Analysis 3: Comparison: Placebo vs Cinacalcet; Test type: Superiority or Other; Difference = 75.44, 95% CI 2-sided [63.83 to 87.05] — Difference = Cinacalcet-Placebo

2. Secondary Outcome: Percent Change From Baseline to Week 52 in Bone Mineral Density at the Femoral Neck
Description: Bone mineral density (BMD) was measured using dual X-ray absorptiometry (DXA).
Time Frame: Baseline and Week 52
Population: Full analysis set with available data
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Placebo | Cinacalcet
Number analyzed (Participants) | 49 | 52
percent change | 1.05 [-1.80 to 3.51] | 1.24 [-1.52 to 4.70]
Statistical Analysis 1: Comparison: Placebo vs Cinacalcet; Test type: Superiority or Other; p = 0.266, ANCOVA; Analysis of covariance (ANCOVA) with Baseline corrected total serum calcium group as a covariate; Difference = 1.41, 95% CI 2-sided [-1.10 to 3.93] — Least square estimate for the difference in the percent change in BMD between the 2 treatment groups (cinacalcet - placebo)

3. Secondary Outcome: Change From Baseline to the EAP in Mean Serum Phosphorus
Time Frame: Baseline and the EAP (mean of Weeks 22, 24, and 26)
Population: Full analysis set with available data
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Cinacalcet
Number analyzed (Participants) | 56 | 56
mg/dL | 0.07 (0.48) | 0.52 (0.54)
Statistical Analysis 1: Comparison: Placebo vs Cinacalcet; Test type: Superiority or Other; p < 0.001, ANCOVA; Analysis of covariance (ANCOVA) with Baseline corrected total serum calcium group as a covariate; Difference = 0.45, 95% CI 2-sided [0.26 to 0.64] — Least square estimate for the difference in the absolute change in mean serum phosphorus between the 2 treatment groups (cinacalcet - placebo)

4. Secondary Outcome: Change From Baseline to Week 52 in eGFR
Description: eGFR was calculated using the Modification of Diet in Renal Disease (MDRD) formula.
Time Frame: Baseline and Week 52
Population: Full analysis set with available data
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m²
Arm/Group | Placebo | Cinacalcet
Number analyzed (Participants) | 52 | 51
mL/min/1.73 m² | 0.06 (8.70) | -0.37 (11.69)
Statistical Analysis 1: Comparison: Placebo vs Cinacalcet; Test type: Superiority or Other; p = 0.842, ANCOVA; ANCOVA with Baseline corrected total serum calcium group as a covariate; Difference = -0.40, 95% CI 2-sided [-4.37 to 3.57] — Least square estimate for the difference in the absolute change in mean eGFR between the 2 treatment groups (cinacalcet - placebo)

5. Secondary Outcome: Change From Baseline to the EAP in Corrected Total Calcium
Time Frame: Baseline and the EAP (mean of Weeks 22, 24, and 26)
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Cinacalcet
Number analyzed (Participants) | 57 | 57
mg/dL | -0.14 (0.51) | -1.53 (0.74)
Statistical Analysis 1: Comparison: Placebo vs Cinacalcet; Test type: Superiority or Other; p < 0.001, ANCOVA; ANCOVA with Baseline corrected total serum calcium group as a covariate; Difference = -1.39, 95% CI 2-sided [-1.62 to -1.16] — Least square estimate for the difference in the absolute change in corrected total calcium between the 2 treatment groups (cinacalcet - placebo)

6. Secondary Outcome: Change From Baseline to the EAP in Intact Parathyroid Hormone (iPTH)
Time Frame: Baseline and the EAP (mean of Weeks 22, 24, and 26)
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo | Cinacalcet
Number analyzed (Participants) | 57 | 57
pg/mL | -10.6 (106.4) | -127.9 (254.2)
Statistical Analysis 1: Comparison: Placebo vs Cinacalcet; Test type: Superiority or Other; p = 0.002, ANCOVA; ANCOVA with Baseline corrected total serum calcium group as a covariate; Difference = -117.21, 95% CI 2-sided [-189.88 to -44.55] — Least square estimate for the difference in the absolute change in iPTH between the 2 treatment groups (cinacalcet - placebo)

7. Secondary Outcome: Change From Baseline to the EAP in Urine Phosphorus
Time Frame: Baseline and the EAP (mean of Weeks 22, 24, and 26)
Population: Full analysis set with available data
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Cinacalcet
Number analyzed (Participants) | 56 | 53
mg/dL | -1.47 (31.51) | -2.62 (43.93)
Statistical Analysis 1: Comparison: Placebo vs Cinacalcet; Test type: Superiority or Other; p = 0.846, ANCOVA; ANCOVA with Baseline corrected total serum calcium group as a covariate; Difference = -1.42, 95% CI 2-sided [-15.91 to 13.06] — Least square estimate for the difference in the absolute change in urine phosphorus between the 2 treatment groups (cinacalcet - placebo)

8. Secondary Outcome: Percentage of Participants With a Parathyroidectomy
Time Frame: 56 weeks
Population: Full analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Cinacalcet
Number analyzed (Participants) | 57 | 57
percentage of participants | 0.0 | 0.0

9. Secondary Outcome: Time to Parathyroidectomy
Time Frame: 56 weeks
Population: Full analysis set who underwent a parathyroidectomy
Arm/Group | Placebo | Cinacalcet
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 60 Weeks
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Placebo | Cinacalcet
Serious Adverse Events (participants affected / at risk) | 19/57 | 15/57
Other Adverse Events (participants affected / at risk) | 45/57 | 45/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=57) | Cinacalcet (N=57)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Glaucoma (Eye disorders) | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Influenza like illness (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Kidney transplant rejection (Immune system disorders) | 0 | 1
Transplant rejection (Immune system disorders) | 1 | 0
Cystitis (Infections and infestations) | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 1 | 2
Escherichia sepsis (Infections and infestations) | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 0 | 1
Muscle abscess (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Urostomy complication (Injury, poisoning and procedural complications) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1
Ureteric stenosis (Renal and urinary disorders) | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 0
Intermittent claudication (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=57) | Cinacalcet (N=57)
Anaemia (Blood and lymphatic system disorders) | 3 | 1
Abdominal discomfort (Gastrointestinal disorders) | 2 | 3
Abdominal pain (Gastrointestinal disorders) | 5 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 8
Nausea (Gastrointestinal disorders) | 6 | 7
Vomiting (Gastrointestinal disorders) | 4 | 3
Fatigue (General disorders) | 7 | 6
Influenza like illness (General disorders) | 3 | 0
Malaise (General disorders) | 0 | 4
Oedema peripheral (General disorders) | 8 | 6
Nasopharyngitis (Infections and infestations) | 8 | 7
Upper respiratory tract infection (Infections and infestations) | 2 | 5
Urinary tract infection (Infections and infestations) | 6 | 8
Decreased appetite (Metabolism and nutrition disorders) | 3 | 2
Gout (Metabolism and nutrition disorders) | 0 | 3
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 | 4
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 3 | 1
Headache (Nervous system disorders) | 3 | 5
Insomnia (Psychiatric disorders) | 1 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 0
Hypertension (Vascular disorders) | 2 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.